CLINICAL TRIAL: NCT06824220
Title: Effect of High-Flow Tracheal Oxygen on End-Expiratory Lung Impedance in Tracheostomized Patients
Brief Title: Effect of High-Flow Tracheal Oxygen on EELI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Argentinian Intensive Care Society (Other)
Responsible Party: Principal Investigator, Gustavo Plotnikow, Hospital Británico de Buenos Aires, Argentinian Intensive Care Society
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: #09122024
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Tracheostomized Patients
Keywords: end-expiratory lung impedance; high-flow tracheal oxygen; Tracheostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- High-Flow Tracheal Oxygen 70 and 80 L/m in Tracheostomized Patients (Other): Implementation of High-Flow Tracheal Oxygen 70 and 80 L/m in Tracheostomized Patients for 20 minutes and End-Expiratory Lung Impedance evaluation
  Interventions: Device: High-Flow Tracheal Oxygen

INTERVENTIONS:
Device: High-Flow Tracheal Oxygen — High-Flow Tracheal Oxygen is the use of high oxygen flows in tracheostomized patients. Unlike conventional oxygen therapy which is performed through siliconized nasal prongs, this is done through a connector directly on the tracheostomy tube.

SUMMARY:
The goal of this analytical experimental study is to evaluate whether high-flow tracheal oxygen therapy at flow rates above 60 L/min increases end-expiratory lung impedance in tracheostomized patients in the intensive care unit. The main question it aims to answer is whether high-flow tracheal oxygen therapy improves end-expiratory lung impedance in tracheostomized patients.

This study will be conducted in the Intensive Care Unit of Sanatorio Parque in Rosario, Santa Fe, Argentina, between December 1, 2024, and March 31, 2025. The participant population consists of adult ICU patients (≥18 years old) who are tracheostomized, have undergone at least 10 days of mechanical ventilation, and can tolerate spontaneous breathing for at least 12 hours.

By analyzing the effects of high-flow tracheal oxygen therapy on lung function, this study aims to generate valuable insights into its physiological impact, potentially influencing clinical management strategies for tracheostomized patients in intensive care settings.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent; ability to tolerate spontaneous breathing for at least 12 hours; arterial oxygen pressure (PaO2) ≥ 60 mm hg or pulse oxygen saturation (SpO2) > 90%; corrected metabolic disorders ph ≥ 7.32; hemodynamically stable.

Exclusion Criteria:

* neuromuscular or neurodegenerative pathology; contraindication for the use of Electrical Impedance Tomography, RASS > +1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
End-Expiratory Lung Impedance | From enrollment to the end of treatment at 120 minutes for each patient
  End-Expiratory Lung Impedance refers to the electrical impedance of lung tissue measured at the end of expiration, serving as a non-invasive indicator of end-expiratory lung volume (EELV). In the context of high-flow oxygen therapy, changes in EELI reflect variations in lung aeration and recruitment in tracheostomized patients.

SECONDARY OUTCOMES:
Respiratory rate | From enrollment to the end of treatment at 120 minutes for each patient
  Respiratory rate refers to the number of breaths a person takes per minute.
Arterial oxygen saturation | From enrollment to the end of treatment at 120 minutes for each patient
  Arterial oxygen saturation refers to the percentage of hemoglobin in the arterial blood that is bound to oxygen. It is a key indicator of oxygenation efficiency and respiratory function

CONTACTS AND LOCATIONS:
Locations (1):
- Sanatorio Parque, Rosario, Santa Fe Province, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Parke RL, Bloch A, McGuinness SP. Effect of Very-High-Flow Nasal Therapy on Airway Pressure and End-Expiratory Lung Impedance in Healthy Volunteers. Respir Care. 2015 Oct;60(10):1397-403. doi: 10.4187/respcare.04028. Epub 2015 Sep 1. PMID 26329355
- [Background] Basile MC, Mauri T, Spinelli E, Dalla Corte F, Montanari G, Marongiu I, Spadaro S, Galazzi A, Grasselli G, Pesenti A. Nasal high flow higher than 60 L/min in patients with acute hypoxemic respiratory failure: a physiological study. Crit Care. 2020 Nov 23;24(1):654. doi: 10.1186/s13054-020-03344-0. PMID 33225971
- [Background] Stripoli T, Spadaro S, Di Mussi R, Volta CA, Trerotoli P, De Carlo F, Iannuzziello R, Sechi F, Pierucci P, Staffieri F, Bruno F, Camporota L, Grasso S. High-flow oxygen therapy in tracheostomized patients at high risk of weaning failure. Ann Intensive Care. 2019 Jan 7;9(1):4. doi: 10.1186/s13613-019-0482-2. PMID 30617626
- [Background] Natalini D, Grieco DL, Santantonio MT, Mincione L, Toni F, Anzellotti GM, Eleuteri D, Di Giannatale P, Antonelli M, Maggiore SM. Physiological effects of high-flow oxygen in tracheostomized patients. Ann Intensive Care. 2019 Oct 7;9(1):114. doi: 10.1186/s13613-019-0591-y. PMID 31591659
- [Background] Corley A, Edwards M, Spooner AJ, Dunster KR, Anstey C, Fraser JF. High-flow oxygen via tracheostomy improves oxygenation in patients weaning from mechanical ventilation: a randomised crossover study. Intensive Care Med. 2017 Mar;43(3):465-467. doi: 10.1007/s00134-016-4634-7. Epub 2016 Nov 30. No abstract available. PMID 27904928
- [Background] Mauri T, Turrini C, Eronia N, Grasselli G, Volta CA, Bellani G, Pesenti A. Physiologic Effects of High-Flow Nasal Cannula in Acute Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2017 May 1;195(9):1207-1215. doi: 10.1164/rccm.201605-0916OC. PMID 27997805
- [Background] Rose L, Messer B. Prolonged Mechanical Ventilation, Weaning, and the Role of Tracheostomy. Crit Care Clin. 2024 Apr;40(2):409-427. doi: 10.1016/j.ccc.2024.01.008. Epub 2024 Feb 2. PMID 38432703
- [Background] Fernandez MM, Gonzalez-Castro A, Magret M, Bouza MT, Ibanez M, Garcia C, Balerdi B, Mas A, Arauzo V, Anon JM, Ruiz F, Ferreres J, Tomas R, Alabert M, Tizon AI, Altaba S, Llamas N, Fernandez R. Reconnection to mechanical ventilation for 1 h after a successful spontaneous breathing trial reduces reintubation in critically ill patients: a multicenter randomized controlled trial. Intensive Care Med. 2017 Nov;43(11):1660-1667. doi: 10.1007/s00134-017-4911-0. Epub 2017 Sep 22. PMID 28936675
- [Background] Navalesi P, Frigerio P, Patzlaff A, Haussermann S, Henseke P, Kubitschek M. Prolonged weaning: from the intensive care unit to home. Rev Port Pneumol. 2014 Sep-Oct;20(5):264-72. doi: 10.1016/j.rppneu.2014.04.006. Epub 2014 Jun 26. PMID 24975297
- [Background] Pham T, Heunks L, Bellani G, Madotto F, Aragao I, Beduneau G, Goligher EC, Grasselli G, Laake JH, Mancebo J, Penuelas O, Piquilloud L, Pesenti A, Wunsch H, van Haren F, Brochard L, Laffey JG; WEAN SAFE Investigators. Weaning from mechanical ventilation in intensive care units across 50 countries (WEAN SAFE): a multicentre, prospective, observational cohort study. Lancet Respir Med. 2023 May;11(5):465-476. doi: 10.1016/S2213-2600(22)00449-0. Epub 2023 Jan 21. PMID 36693401
- [Background] Mussa CC, Gomaa D, Rowley DD, Schmidt U, Ginier E, Strickland SL. AARC Clinical Practice Guideline: Management of Adult Patients with Tracheostomy in the Acute Care Setting. Respir Care. 2021 Jan;66(1):156-169. doi: 10.4187/respcare.08206. Epub 2020 Sep 22. PMID 32962998